CLINICAL TRIAL: NCT06001450
Title: PLANET: Exploring the Role of Plastics and Toxins in Intestinal Inflammation
Brief Title: Pregnant Women With and Without Crohns Disease to Explore the Role of Plastics and Toxins in Intestinal Inflammation
Acronym: PLANET
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Manasi Agrawal, Assistant Professor of Medicine, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-23-00245; 22-1179-00001 (Other Grant/Funding Number: Crohn's & Colitis Foundation Of America)
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-10

CONDITIONS: Crohns Disease; Pregnancy; Inflammatory Bowel Disease
Keywords: microplastics; nanoplastics; pregnancy; pollution; environmental pollutants
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool, Saliva, Breast milk, Whole Blood (optional), Cord Blood (optional), Placenta (optional)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pregnant people with Crohns disease (Case): Arm 1 is pregnant people with Crohns disease who enroll with the infant that they are pregnant with at the time.
- Pregnant people without Crohns disease (Control): Arm 2 is the control arm of pregnant people without Crohns disease and other inflammatory bowel diseases who enroll with the infant that they are pregnant with at the time.

SUMMARY:
The PLANET Study aims to determine the impact of microplastics on intestinal inflammation and gut microbiome in order to understand the role of this pollutant on the risk of developing inflammatory bowel disease (IBD) as well as other diseases. With this information, the researchers hope to characterize better the role of environmental pollutants on IBD and develop novel strategies towards prevention.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD), including Crohn's disease (CD) and ulcerative colitis (UC), is a chronic, progressive inflammatory disease of the intestinal tract. The etiology of IBD is not well understood, but believed to result from a complex relationship between genetics, environment, and gut microbiome alterations, resulting in a self-perpetuating, abnormal mucosal immune response. The incidence of IBD is rising in developing and recently developed countries, highlighting the importance of environmental exposures in determining disease risk. Microplastics, defined as plastic particles <5 mm in size, are ubiquitous pollutants with unclear implications towards human health. Emerging studies indicate substantial disruption of intestinal immune function and a proinflammatory milieu due to microplastics. Therefore, identifying, and characterizing microplastics in stool samples of individuals with CD alongside alterations in microbiome and calprotectin, which are events that occur prior to CD onset, is the initial step in exploring the impact of microplastics on IBD. Moreover, CD affects women during their reproductive years and 25% become pregnant after diagnosis. Given that maternal IBD diagnosis is one of the major risks of future IBD in offspring, it is critical to better understand if babies born to mothers with IBD have higher content of microplastics or other toxins in the stools and whether these levels correlate with those of their mothers during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* The ability to sign and date an informed consent form
* Be pregnant, or wishing to become pregnant in the near future and enroll the infant that the individual is pregnant with
* Aged 18 or older
* English-speaking (this observational study uses non-validated questionnaires that are only available in English)
* Of any ethnicity
* Be a spouse, related household member (sibling, parent, etc.) or a child of an enrolled pregnant person

Exclusion Criteria:

* Individuals who are unable to give informed consent
* Be diagnosed with a pregnancy complication, such as intrauterine fetal demise/stillbirth, preeclampsia, hyperemesis gravidarum, or have an active infection, including chorioamnionitis or sepsis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant people 18 years and older, with and without Crohns disease.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Microplastics quantification | 1 year
  Measuring the concentration, size and shape distributions of microplastics in the stool samples of women with CD, healthy controls and any relatives (spouses and siblings of the infant).

SECONDARY OUTCOMES:
Alpha and beta diversity | 1 year
  Microbiome characterization - Bacterial DNA will be isolated from stool and sequenced to characterize the bacteria present in the microbiome. Alpha and beta diversity statistics will be reported.
Fecal calprotectin analysis | 1 year
  Stool samples will be processed to quantify calprotectin levels which are routinely used to characterize inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Manasi Agrawal, MD, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no blanket statement on IPD as some participants may opt out of data sharing in collaborations and the researchers will not be submitting data to any repositories.